CLINICAL TRIAL: NCT00420355
Title: The Pharmacokinetics of Lopinavir/Ritonavir in Combination With Atazanavir in HIV-Infected Subjects
Brief Title: Pharmacokinetic Study of Two HIV Protease Inhibitors in Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unexpected adverse event
Sponsor: University of Oklahoma (Other)
Collaborators: Abbott (Industry)
Responsible Party: R. Chris Rathbun, Pharm.D., University of Oklahoma Health Sciences Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12637
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infection
Keywords: antiretroviral therapy; protease inhibitors; drug interactions; HIV infection; acquired immunodeficiency syndrome; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Subjects on atazanavir/ritonavir will add lopinavir/ritonavir.
  Interventions: Drug: lopinavir/ritonavir
- Arm B (Experimental): Subjects on lopinavir/ritonavir will add atazanavir.
  Interventions: Drug: atazanavir

INTERVENTIONS:
Drug: atazanavir — Atazanavir 300 mg daily on Days 6-12.
  Other Names: Reyataz 300 mg capsules
  Arms: Arm B
Drug: lopinavir/ritonavir — Lopinavir/ritonavir 400 mg/100 mg twice daily on Days 6-16, then 800 mg/200 mg daily on Days 17-21.
  Other Names: Kaletra 200 mg/50 mg tablets
  Arms: Arm A

SUMMARY:
The objective of this study is to determine the pharmacokinetics of lopinavir, ritonavir, and atazanavir when lopinavir/ritonavir and atazanavir are used in combination.

DETAILED DESCRIPTION:
Thirty patients with HIV infection will be enrolled in this open-label, parallel arm pharmacokinetic study. Subjects receiving either lopinavir/ritonavir or atazanavir/ritonavir as part of their antiretroviral therapy will have a pharmacokinetic study performed over 12-20 days to examine whether coadministration of lopinavir and atazanavir alters the pharmacokinetics of either agent. The safety of these agents in combination will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* HIV-seropositive
* Currently receiving atazanavir/ritonavir or lopinavir/ritonavir in combination with 2-3 nucleoside RT inhibitors or are antiretroviral treatment-naïve
* If female, is not of childbearing potential or is of childbearing potential and agrees to use a barrier method of contraception throughout the study

Exclusion Criteria:

* HIV-1 RNA > 400 copies/mL if currently receiving antiretroviral therapy
* Concurrent use of CYP450 inhibitors or inducers
* Concurrent use of P-glycoprotein substrates, inhibitors, or inducers
* Concurrent use of medications known to interact with ritonavir or atazanavir
* Presence of a chronic health condition deemed by the investigators to potentially impair lopinavir, ritonavir, or atazanavir pharmacokinetics
* Presence of conduction abnormalities on electrocardiogram
* Women who are pregnant or breastfeeding
* Laboratory Abnormalities at baseline:

  * Aminotransferases > 3x ULN
  * Serum bilirubin > 5x ULN
  * Serum creatinine > 1.5x ULN
  * Hemoglobin concentration < 8.0 g/dL
  * Absolute neutrophil count < 800 cells/μL
  * Platelet count < 50,000 cells/μL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Mean pharmacokinetic parameters (Cmax, Cmin, AUC) for lopinavir, ritonavir, atazanavir | Day 6, Day 12 or 16, Day 20

SECONDARY OUTCOMES:
Safety (e.g., GI tolerance, lab abnormalities, ECG changes) | Day 6, Day 12 or Day 16, Day 20

CONTACTS AND LOCATIONS:
Overall Officials: R. Chris Rathbun, Pharm.D., Principal Investigator — University of Oklahoma
Locations (1):
- OUHSC General Clinical Research Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Rathbun CR, Liedtke MD, Blevins SM, Harrison D, Lockhart SM, Salvaggio M, Acosta EP. Electrocardiogram abnormalities with atazanavir and lopinavir/ritonavir. HIV Clin Trials. 2009 Sep-Oct;10(5):328-36. doi: 10.1310/hct1005-328. PMID 19906626